CLINICAL TRIAL: NCT03079921
Title: Adrenergic Contribution to Glucose Counterregulation in Islet Transplantation
Brief Title: Adrenergic System in Islet Transplantation
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael R. Rickels, MD, MS, Michael R. Rickels, M.D., M.S. Associate Professor of Medicine Division of Endocrinology, Diabetes & Metabolism Director, Translational Research Program Institute for Diabetes, Obesity & Metabolism University of Pennsylvania Perelman School of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 826386; 2R01DK091331-06 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-15 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Type1diabetes; Hypoglycemia; Hypoglycemia Unawareness; Islet Cell Transplantation
Keywords: Islet Graft Function; Islet Cell transplantation; Auto-islet transplantation; Intra-hepatic islets; Extra-hepatic islets
MeSH Terms: conditions — Hypoglycemia | interventions — Phentolamine; Propranolol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study is a within subject and across group mechanistic design.
  Islet cell hormonal responses to a hyperinsulinemic euglycemic-hypoglycemic clamp will be assessed in "Group 1" on three occasions with randomized, double-blind administration of the α-adrenergic blocker phentolamine, the β-adrenergic blocker propranolol, or placebo.
  Responses in "Group 1" under the placebo condition will be used for comparison to those obtained from hyperinsulinemic euglycemic-hypoglycemic clamp testing on one occasion in subjects in each of "Group 2" and "Group 3".
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Conditions of testing for "Group 1" (intra-hepatic islet recipients) will remain double-blind for each subject until their completion of all testing visits, unless for safety concerns, either the PI or Medical Monitor request an unblinding. Groups "2" and "3" will have no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1-Propranolol Intra-hepatic islet (Active Comparator): The dose of propranolol will be 0.48 μg/kilogram•minute, which will provide a total dose of 0.10 mg/kg. It will be administered 1 x only via intravenous infusion over 3.5 hours, starting 30 min before conduct of a hyperinsulinemic euglycemic (90 min) followed by hypoglycemia (90 min) clamp.
  Interventions: Drug: Propranolol
- Group 1-Phentolamine Intra-hepatic islet (Active Comparator): The dose of phentolamine will be 0.95 μg/kg•min, which will provide a total dose of 0.20 mg/kg. It will be administered 1 x only via intravenous infusion over 3.5 hours, starting 30 min before conduct of a hyperinsulinemic euglycemic (90 min) followed by hypoglycemia (90 min) clamp.
  Interventions: Drug: Phentolamine
- Group 1- Placebo Intra-hepatic islet (Placebo Comparator): Placebo in 100mL NSS. Infuse Intravenously at 0.0095 ML/KG/MIN. 1 x only via intravenous infusion over 3.5 hours, starting 30 min before conduct of a hyperinsulinemic euglycemic (90 min) followed by hypoglycemia (90 min) clamp.
  Interventions: Drug: Placebo
- Group 2 - Extra-hepatic islet (No Intervention): Hyperinsulinemic euglycemic (90 min) followed by hypoglycemia (90 min) clamp only.
- Group 3 - Intra-hepatic auto islet (No Intervention): Hyperinsulinemic euglycemic (90 min) followed by hypoglycemia (90 min) clamp only.

INTERVENTIONS:
Drug: Phentolamine — Physiologic receptor blockade (α1-receptor).
  Other Names: Regitine
  Arms: Group 1-Phentolamine Intra-hepatic islet
Drug: Propranolol — Physiologic receptor blockade (β2-receptor).
  Other Names: Inderal
  Arms: Group 1-Propranolol Intra-hepatic islet
Drug: Placebo — 100mL bag of Normal Saline Solution (NSS).
  Other Names: Saline; Sodium Chloride Solution
  Arms: Group 1- Placebo Intra-hepatic islet

SUMMARY:
To determine the effect of sympathetic neural and hormonal (epinephrine) input on islet cell hormonal responses to insulin-induced hypoglycemia in type 1 diabetic recipients of intrahepatic islet transplantation. We hypothesize that α-adrenergic (neural) blockage will abolish insulin-mediated suppression of C-peptide, attenuating α-cell glucagon secretion during hypoglycemia, and that β-adrenergic (hormonal) blockage will have no effect. Glucose counterregulatory responses will be measured during hyperinsulinemic euglycemic-hypoglycemic clamps on three occasions with randomized, double-blind administration of the α-adrenergic blocker phentolamine, the β-adrenergic blocker propranolol, or placebo. The demonstration of neural rather than hormonal regulation of the transplanted islet cell response to hypoglycemia is critical for understanding the mechanism for protection from hypoglycemia afforded by intrahepatically transplanted.

DETAILED DESCRIPTION:
This study is designed to test the hypothesis that α-adrenergic (neural) blockade will abolish insulin-mediated suppression of C-peptide, attenuating α-cell glucagon secretion during hypoglycemia, and that β-adrenergic (hormonal) blockade will have no effect. Glucose counterregulatory responses will be measured during hyperinsulinemic euglycemic-hypoglycemic clamps on three occasions with randomized, double-blind administration of the α-adrenergic blocker phentolamine, the β-adrenergic blocker propranolol, or placebo. The demonstration of neural rather than hormonal regulation of the transplanted islet cell response to hypoglycemia is critical for understanding the mechanism for protection from hypoglycemia afforded by intrahepatically transplanted islets.

Glucose counterregulation has not been studied in type 1 diabetic recipients of extrahepatic islet transplantation. Comparison of glucose counterregulatory responses measured during hyperinsulinemic euglycemic-hypoglycemic clamps will be compared to those obtained from type 1 diabetic recipients of intrahepatic islet transplantation studied under the placebo condition above.

Glucose counterregulation has not been directly compared between recipients of intrahepatic auto- and allo-islet transplantation. Direct comparison of glucose counterregulatory responses under the same experimental conditions is required to understand whether mechanisms other than the glucagon response may be important to the reported hypoglycemia affecting pancreatectomized recipients of islet auto-transplantation.

ELIGIBILITY:
Inclusion Criteria:

GROUP 1

1. Male and female subjects age 21 to 65 years of age.
2. Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
3. Clinical history compatible with type 1 diabetes with onset of disease at < 40 years of age and insulin-dependent for > 10 years at the time of islet transplantation > 6 months before study.
4. Stable islet graft function defined by C-peptide > 0.5 ng/ml and insulin-independent or insulin-dependent with daily insulin requirement < 0.2 units/kg•d to maintain HbA1c < 7.0%.
5. Use of standard immunosuppression consisting of tacrolimus with or without sirolimus or mycophenolic acid. Substitutions of tacrolimus with cyclosporine, and of sirolimus or mycophenolic acid with azathioprine are permissible if stable for over 3 months. Prednisone is allowable if no more than 5 mg daily.

Exclusion Criteria:

GROUP 1

1. BMI ≥ 30 kg/m2.
2. Insulin requirement of ≥ 0.2 units/kg•day.
3. HbA1c ≥ 7.0%.
4. Uncontrolled hypertension: systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
5. History of cardiovascular disease, including coronary artery, cerebrovascular or peripheral vascular disease, or current use of β-blocker therapy.
6. Bronchial asthma.
7. Abnormal kidney function: Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2.
8. Abnormal liver function: persistent elevation of liver function tests > 1.5 times the upper limit of normal.
9. Untreated hypothyroidism, Addison's disease, or Celiac disease.
10. Anemia: baseline hemoglobin concentration < 11 g/dl in women and < 12 g/dl in men.
11. Presence of a seizure disorder not related to prior severe hypoglycemia.
12. Use of glucocorticoids greater than 5 mg of prednisone daily, or an equivalent physiologic dose of hydrocortisone.
13. For female participants of child-bearing potential: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of study participation. Oral contraceptives, intra-uterine devices, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
14. Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment.
15. Use of any investigational agents within 4 weeks of enrollment.
16. Any medical condition that, in the opinion of the PI, will interfere with the safe completion of the study

Inclusion Criteria GROUP 2

1. Male and female subjects age 21 to 65 years of age.
2. Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
3. Clinical history compatible with type 1 diabetes with onset of disease at < 40 years of age and insulin-dependent for > 10 years at the time of islet transplantation > 6 months before study.
4. Stable islet graft function defined by C-peptide > 0.5 ng/ml and insulin-independent or insulin-dependent with daily insulin requirement < 0.2 units/kg•d to maintain HbA1c < 7.0%.
5. Use of standard immunosuppression consisting of tacrolimus with or without sirolimus or mycophenolic acid. Substitutions of tacrolimus with cyclosporine, and of sirolimus or mycophenolic acid with azathioprine are permissible if stable for over 3 months. Prednisone is allowable if no more than 5 mg daily.

Exclusion Criteria:

GROUP 2

1. BMI ≥ 30 kg/m2.
2. Insulin requirement of ≥ 0.2 units/kg•day.
3. HbA1c ≥ 7.0%.
4. Uncontrolled hypertension: systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
5. Active cardiovascular disease, including coronary artery, cerebrovascular or peripheral vascular disease.
6. Abnormal kidney function: eGFR < 60 ml/min/1.73 m2.
7. Abnormal liver function: persistent elevation of liver function tests > 1.5 times the upper limit of normal.
8. Untreated hypothyroidism, Addison's disease, or Celiac disease.
9. Anemia: baseline hemoglobin concentration < 11 g/dl in women and < 12 g/dl in men.
10. Presence of a seizure disorder not related to prior severe hypoglycemia.
11. Use of glucocorticoids greater than 5 mg of prednisone daily, or an equivalent physiologic dose of hydrocortisone.
12. For female participants of child-bearing potential: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of study participation. Oral contraceptives, intra-uterine devices, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
13. Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment.
14. Use of any investigational agents within 4 weeks of enrollment.
15. Any medical condition that, in the opinion of the PI, will interfere with the safe completion of the study

Inclusion Criteria GROUP 3

Patients who meet all of the following criteria are eligible for participation in Group 3 of this study:

1. Male and female subjects age 21 to 65 years of age.
2. Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
3. Clinical history compatible with total pancreatectomy and autologous islet transplantation > 6 months before study.
4. Stable islet graft function defined by C-peptide > 0.5 ng/ml and insulin-independent or insulin-dependent with daily insulin requirement < 0.2 units/kg•d to maintain HbA1c < 7.0%.

Exclusion Criteria:

GROUP 3

1. BMI ≥ 30 kg/m2.
2. Insulin requirement of ≥ 0.2 units/kg•day.
3. HbA1c ≥ 7.0%.
4. Uncontrolled hypertension: systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
5. Active cardiovascular disease, including coronary artery, cerebrovascular or peripheral vascular disease.
6. Abnormal kidney function: eGFR < 60 ml/min/1.73 m2.
7. Abnormal liver function: persistent elevation of liver function tests > 1.5 times the upper limit of normal.
8. Anemia: baseline hemoglobin concentration < 11 g/dl in women and < 12 g/dl in men.
9. Presence of a seizure disorder not related to prior severe hypoglycemia.
10. Use of glucocorticoids greater than 5 mg of prednisone daily, or an equivalent physiologic dose of hydrocortisone.
11. For female participants of child-bearing potential: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of study participation. Oral contraceptives, intra-uterine devices, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
12. Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment.
13. Use of any investigational agents within 4 weeks of enrollment.
14. Any medical condition that, in the opinion of the PI, will interfere with the safe completion of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or Female at birth.
Enrollment: 11 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
C-PEPTIDE suppression during hyperinsulinemia euglycemia. | For C-peptide at the 60-90 time-point during the hyperinsulinemic euglycemic-hypoglycemic clamp.
  The primary outcome measures will be the levels of C-peptide during hyperinsulinemia euglycemia.
GLUCAGON activation during hyperinsulinemia hypoglycemia. | For Glucagon at the 150-180 minute time-point during the hyperinsulinemic euglycemic-hypoglycemic clamp.
  The primary outcome measures will be the levels of glucagon during hyperinsulinemia hypoglycemia.

SECONDARY OUTCOMES:
EPINEPHRINE during hyperinsulinemia hypoglycemia. | During metabolic testing in the 150-180 minute time-point of the hyperinsulinemic euglycemic-hypoglycemic clamp.
  Secondary outcome measures will include levels of epinephrine during hyperinsulinemia hypoglycemia.
Rates of ENDOGENOUS GLUCOSE PRODUCTION during hyperinsulinemia hypoglycemia. | During metabolic testing in the 150-180 minute time-point of the hyperinsulinemic euglycemic-hypoglycemic clamp.
  Secondary outcome measures will include rates of endogenous glucose production during hyperinsulinemia hypoglycemia
AUTONOMIC SYMPTOMS during hyperinsulinemia | During metabolic testing; this symptom questionnaire will be asked at the following time points: -15min, -1min, 30min, 60min,75min, 90min,120min, 150min, 165min, 180min.
  Secondary outcome measures will include levels of autonomic symptoms during hyperinsulinemia hypoglycemia. Autonomic symptoms will be measured by answering a short symptoms questionnaire with a level scale of 0-5.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Rickels, MD., MS, Principal Investigator — Division of Endocrinology, Diabetes & Metabolism, Perelman School of Medicine
Locations (1):
- University of Pennsylvania - Institute for Diabetes, Obesity and Metabolism, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be any further plan to make IPD available besides the Informed Consent.

REFERENCES:
- See also: Perelman School of Medicine / Faculty Search /Michael Rickels, M.D., M.S. — https://www.med.upenn.edu/apps/faculty/index.php/p32032
- See also: Research Studies at the University of Pennsylvania — https://clinicalresearch.itmat.upenn.edu/?_ga=1.86091032.1687586810.1437483178
- See also: Institute for Diabetes, Obesity and Metabolism Research Studies — https://www.med.upenn.edu/idom/trials.html

DOCUMENTS (1):
  • Informed Consent Form (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT03079921/ICF_000.pdf